CLINICAL TRIAL: NCT00581906
Title: Dynamic Contrast Enhanced MRI (DCE-MRI) Diffusion Weighted MRI (DW-MRI) and Magnetic Resonance Spectroscopy (MRS) of Head and Neck Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 06-007; NIH R01 CA115895
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Head Cancer; Neck Cancer; Dynamic Contrast Enhanced MRI; Magnetic Resonance Spectroscopy (MRS); Diffusion Weighted MRI (DW-MRI); 06-007
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- pts undergoing surgery or chemo-radiation treatment
  Interventions: Radiation: DCE-MRI, DW-MRI and MRS

INTERVENTIONS:
Radiation: DCE-MRI, DW-MRI and MRS — Pts undergo DCE-MRI, DW-MRI or 1^H-MRS studies on either the 1.5T scanner or the 3T MRI scanners. Patients will be grouped based on their treatment: group one will include pts who undergo surgery (we will no longer accrue pts in this group) & group two will include pts who undergo chemoradiation therapy.Pts who undergo surgery will have pretreatment DCE-MRI, DW-MRI &/or 1H-MRS studies on the GE 1.5T or 3T MRI scanner. Pts who participate in chemo-radiation therapy protocols will have pretreatment DCE-MRI, DW-MRI &/or 1H-MRS studies on the 3T Philips MRI scanner in the radiation oncology suite & will undergo additional recommended weekly DW-MRI including IVIM studies at the same MRI scanner during the course of treatment. Pts will undergo two recommended DCE-MRI studies (unless contraindicated) when possible. 1st intra-treatment DCE-MRI is recommended between the 1st & 2nd weeks of treatment & the 2nd intra-treatment DCE-MRI is recommended between the 3rd & 4th weeks of treatment.

SUMMARY:
Magnetic resonance imaging (MRI) is a diagnostic study that makes pictures of organs of the body using magnetic field and radio frequency pulses that can not be felt. Dynamic contrast enhanced-magnetic resonance imaging (DCE-MRI) uses faster imaging and contrast material (a substance used to make specific organs, blood vessels, or tumors easier to see) that is given by vein. Diffusion weighted magnetic resonance imaging (DW-MRI) allows to measure the motion of water around the cells in the tumor. Proton magnetic resonance spectroscopy (MRS) obtains chemical information from the tumor. During MRS, signals are detected from the chemicals (spectroscopy) naturally present in your tumor using radio waves. DCE-MRI, DW-MRI and MRS give extra information which is not available with the regular MRI. The regular MRI only shows pictures of the tumor while the DCE-MRI also gives information about the blood vessels of the tumor. DW-MRI provides information related to the state of the tumor tissue with regards to the quality or condition of cells present in it and MRS gives information about the chemical makeup of the tumor.

The purpose of this study is to see whether DCE-MRI, DW-MRI and MRS done before treatment can predict which patients will do well with either surgery or chemo-radiation therapy. This study will also see if DCE-MRI, DW-MRI and MRS done early in treatment can tell if the therapy is working.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven diagnosis of head and neck cancer or patients with tumors strongly suspicious for head and neck cancer due to clinical features or FNA (fine needle aspiration) cytology assessment.
* Will undergo surgery or chemo-radiation treatment
* Patients must be 18 years or older and have the ability to give informed consent

Exclusion Criteria:

* Claustrophobia
* Known reaction to Gd-DTPA
* Pre-operative radiation to primary tumor site
* Contraindication to MRI

  1. Pacemaker
  2. Aneurysmal clips
  3. Metal implants in field of view
  4. Pregnant or nursing women
  5. Age and mental status wherein he/she is unable to cooperate for MRI study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2006-02; Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Identify a priori prognostic markers for head and neck cancer patients using DCE-MRI, DW-MRI and 1H-MRS data, which may help in stratifying patients into "good risk" and "poor risk" categories to improve outcome and quality of life. | 5 years

SECONDARY OUTCOMES:
To determine if the a-priori DCE-MRI, DW-MRI and 1H-MRS results provide independent markers of tumor response and/or long term disease-free survival compared to clinical prognosticators. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amita Dave, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center website — http://www.mskcc.org

DOCUMENTS (1):
  • Informed Consent Form (2018-05-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT00581906/ICF_000.pdf